CLINICAL TRIAL: NCT03727451
Title: A Dose Escalation Study to Assess the Safety and Efficacy of Pulsed, Inhaled Nitric Oxide in Subjects With Pulmonary Hypertension Associated With Pulmonary Fibrosis or Sarcoidosis on Long Term Oxygen Therapy Followed by an Optional Open-Label Long Term Extension Safety Study
Brief Title: A Dose Escalation Study to Assess the Safety and Efficacy of Pulsed Inhaled Nitric Oxide in Subjects With Pulmonary Fibrosis or Sarcoidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bellerophon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PULSE-PHPF-002
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Hypertension; Pulmonary Fibrosis; Sarcoidosis, Pulmonary
Keywords: Pulmonary Hypertension; Pulmonary Fibrosis; Sarcoidosis
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Fibrosis; Sarcoidosis, Pulmonary; Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PH-Pulmonary Fibrosis (Experimental): Part 1: 1st 4 subjects will be treated with iNO 30, 45, 75 mcg/kg IBW/hr
  2nd 4 subjects will be treated with iNO 45, 75, 125 mcg/kg IBW/hr
  Part 2: Optional open label long term extension at the optimal dose as identified in Part 1
  Interventions: Combination Product: iNO
- PH-Sarcoidosis (Experimental): Part 1: 1st 4 subjects will be treated with iNO 30, 45, 75 mcg/kg IBW/hr
  2nd 4 subjects will be treated with iNO 45, 75, 125 mcg/kg IBW/hr
  Part 2: Optional Open label long term extension at the optimal dose as identified in Part 1
  Interventions: Combination Product: iNO

INTERVENTIONS:
Combination Product: iNO — inhaled nitric oxide
  Other Names: iNOPulse

SUMMARY:
A phase 2b, open label study to assess the safety and efficacy of increasing doses of pulsed, inhaled nitric oxide (iNO) in subjects with pulmonary fibrosis and sarcoidosis on long term oxygen therapy followed by a long term extension study

DETAILED DESCRIPTION:
A phase 2b, open label study to assess the hemodynamic effects of increasing doses of pulsed, inhaled nitric oxide (iNO) in subjects with pulmonary hypertension associated with pulmonary fibrosis or sarcoidosis on long term oxygen therapy followed by an open label extension study

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. A primary diagnosis of sarcoidosis as defined by the ATS/ERS/WASOG statement or pulmonary fibrosis associated with one of the following conditions:

   2.1 Major IIPs (idiopathic interstitial pneumonias) diagnosed or suspected as one of the following:
   * Idiopathic pulmonary fibrosis
   * Idiopathic nonspecific interstitial pneumonia
   * Respiratory bronchiolitis-interstitial lung disease
   * Desquamative interstitial pneumonia
   * Cryptogenic organizing pneumonia
   * Acute interstitial pneumonia
   * Rare IIPs diagnosis by one of the following:
   * Idiopathic lymphoid interstitial pneumonia
   * Idiopathic pleuroparenchymal fibroelastosis
   * Unclassifiable idiopathic interstitial pneumonias

   2.2 Chronic hypersensitivity pneumonitis

   2.3 Occupational lung disease

   2.4 Connective tissue disease with evidence of significant pulmonary fibrosis
3. Intermediate or high probability of PH by echocardiogram as assessed by local Radiologist/Investigator, or PH as determined by a right heart catheterization (RHC) within 5 years prior to Baseline with the following parameters:

   1. Pulmonary vascular resistance (PVR) ˃3 Wood Units (WU) (320 dynes.sec.cm-5)
   2. A left ventricular end diastolic pressure (LVEDP) or pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg
   3. A mean pulmonary arterial pressure (mPAP) of ≥ 25 mmHg
4. 6MWD ≥ 100 meters and ≤ 450 meters
5. WHO Functional Class II-IV
6. Forced Vital Capacity ≥ 40% predicted within last 6 weeks prior to screening
7. Females of childbearing potential must have a negative pre-treatment pregnancy test (urine).
8. Age between 18 and 85 years (inclusive)
9. Clinically stable for at least 4 weeks prior to Baseline in the opinion of the Investigator
10. If on therapy for their parenchymal lung disease and/or sarcoidosis, then the subject should be on a stable well-tolerated dose of the medication(s) for at least 4 weeks prior to enrollment.

Exclusion Criteria:

1. Use of any type of PAH specific therapies
2. Episodes of disease worsening within 3 months prior to Baseline
3. Pregnant or breastfeeding females at Screening
4. Administered L-arginine within 1 month prior to Screening
5. Any subject who has been enrolled in any previous clinical study with inhaled NO administered through pulsed delivery
6. On more than 6 L/min of oxygen at rest by nasal cannula for less than 4 weeks
7. Evidence of any connective tissue disease with FVC > 60% in the last 6 months prior to screening unless there is evidence of moderate to severe fibrosis on CT scan in the opinion of the local radiologist/Investigator
8. Evidence of clinically significant combined pulmonary fibrosis with emphysema (CPFE) if > 15% of lung fields by CT scan show evidence of emphysema in the opinion of the local radiologist/Investigator
9. For subjects with sarcoidosis, clinically significant evidence of pulmonary fibrosis on CT scan in the opinion of the local radiologist/Investigator and FVC ≥80% predicted
10. For subjects continuing on open label therapy, the concurrent use of the INOpulse device with a CPAP/BiPAP, or any other positive pressure device
11. Significant heart failure in the opinion of the Investigator

    1. LVEF<40% or
    2. PCWP on last RHC>15 mmHg (unless concurrent LVEDP <15 mmHg) or
    3. Significant diastolic dysfunction on echocardiogram

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Measurement of mean PAP | During a single right heart catheterization procedure
  Mean pulmonary arterial pressure (mPAP) will be measured at iNO 30, 45, 75 and 125 mcg/kg IBW/hr
Measurement of PCWP | During a single right heart catheterization procedure
  Pulmonary capillary wedge pressure (PCWP) will be measured at iNO 30, 45, 75 and 125 mcg/kg IBW/hr
Measurement of PVR | During a single right heart catheterization procedure
  Pulmonary vascular resistance (PVR) will be measured at iNO 30, 45, 75 and 125 mcg/kg IBW/hr
Measurement of CO | During a single right heart catheterization procedure
  Cardiac output (CO) will be measured at iNO 30, 45, 75 and 125 mcg/kg IBW/hr
Change in 6MWD from Baseline to 16 Weeks | 16 weeks
  Change in 6 minute walk distance

SECONDARY OUTCOMES:
Incidence and Severity of Treatment Emergent Adverse Events | During a single right heart catheterization procedure
  Including adverse events related to device deficiency
Pulmonary Rebound | During a single right heart catheterization procedure
  Symptoms associated with acute withdrawal of iNO: systemic arterial oxygen desaturation, hypoxemia, bradycardia, tachycardia, systemic hypotension, shortness of breath, near-syncope and syncope
Distance Saturation Product (DSP) | 16 weeks
  Difference in DSP from baseline to Week 16
  Difference in DSP from baseline to 16 weeks
Dyspnea | 16 weeks
  Difference in dyspnea as measured by UCSD Medical Center Pulmonary Rehabilitation Program Shortness of Breath Questionnaire on a scale from 0 (none at all) to 5 (maximal or unable to do because of breathlessness) from baseline to Week 16
Quality of Life Assessment | 16 weeks
  Difference in disease specific Quality of Life as measured by St. George's Respiratory Questionnaire
Incidence of Adverse Events and Serious Averse Events | Through study completion; an average of 1 year
  Evaluation of adverse events and serious adverse events
Integral Distance Saturation Product (IDSP) | 16 weeks
  Difference in IDSP from baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Edward Parsley, DO, Study Director — Bellerophon Pulse Technologies
Locations (6):
- United States (6):
  - University of Miami, Miami, Florida
  - University of Cincinnati, Cincinnati, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inova Heart and Lung Vascular Institute, Falls Church, Virginia
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No